CLINICAL TRIAL: NCT02906904
Title: Objective Measures of Pain Sensitivity in NREM Sleep Parasomnia
Brief Title: Pain Sensitivity in NREM Parasomnia (NOCISOMNIE)
Acronym: NOCISOMNIE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Material needed for study was not available
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9540
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: NREM Parasomnia; Sleepwalking; Sleep Terror
MeSH Terms: conditions — Somnambulism; Night Terrors

ARMS (2):
- CASE (adult sleepwalking patients) (Experimental)
  Interventions: Other: Case Intervention
- CONTROL (adult healthy volunteers) (Experimental)
  Interventions: Other: Control Intervention

INTERVENTIONS:
Other: Case Intervention — 24-hour sleep deprivation protocol, polysomnographic monitoring of the recovery sleep, triggering of parasomniac episodes by auditory stimulations, thermoalgic stimulation (Modulator Sensory Analyzer Thermal Stimulator®) during wakefulness, parasomniac episodes, NREM stage 2 ans SWS
  Arms: CASE (adult sleepwalking patients)
Other: Control Intervention — 24-hour sleep deprivation protocol, polysomnographic monitoring of the recovery sleep, thermoalgic stimulation (Modulator Sensory Analyzer Thermal Stimulator®) during wakefulness, NREM stage 2 ans SWS
  Arms: CONTROL (adult healthy volunteers)

SUMMARY:
Non Rapid Eye Movement (NREM) sleep parasomnias (sleepwalking and sleep terrors) are frequent and disabling sleep disorders characterized by arousal specifically from slow wave sleep (SWS) with dissociated brain activity that may be related to lower nociceptive state. The investigators recently reported frequent subjective complaints of chronic pain, migraine and headache during wakefulness in adult sleepwalkers. They also described frequent analgesia during severe and injuring episodes, suggesting a relationship between dissociated brain activity and nociceptive dysregulation. However, this study did not included objective nociceptive measures and the retrospective assessment of perceived pain during parasomnia episodes over a lifetime span might also introduce a recall bias.

The aims of the present study are to measure objective pain sensitivity in patients with NREM parasomnias and matched controls during 1) parasomniac episodes, 2) light NREM sleep and SWS, and 3) wakefulness.

Fifteen adults with severe NREM parasomnia and 15 age and sex-matched controls will be recruited. A 25 hours (8 AM to 9 AM) sleep deprivation protocol followed by auditory stimulations during SWS will be used to trigger parasomniac episodes. Thermoalgic stimulations of graduate intensity will be applied during wakefulness (8 PM) to determine the nociceptive threshold. During the recovery sleep following the sleep deprivation, the investigators will apply repeated subthreshold thermoalgic stimulations in NREM stage 2, SWS and triggered parasomniac episodes and report the behavioural/neurophysiologic nociceptive responses.

The investigators hypothesized a lower nociceptive threshold during wakefulness in sleepwalkers and a decrease of the arousabiliy during SWS and parasomniac episodes. This study may help to better understand the etiology and mechanisms underlying the clinical enigma of the nociceptive dysregulation in NREM sleep parasomnias.

ELIGIBILITY:
Inclusion Criteria:

* Subject from 18 years-old to 45 years-old
* Affiliated to social security
* Written informed consent

  * CASE specific inclusion criteria :
* NREM parasomnia diagnosed according to the International Classification of Sleep Disorders 3rd edition (ICSD-3) criteria and confirmed by polysomnography assessment
* Frequent symptomatology (at least 1 episode by week in the past 3 months)

  * CONTROL specific inclusion criteria :
* No medical history of NREM parasomnia

Exclusion Criteria:

* Known skin allergy to metal
* Use of psychotropic drugs during the 15 days before the inclusion
* Use of analgesic drugs during the 15 days before the inclusion
* A diagnosis of sleep apnea syndrome, periodic limb movements or restless legs syndrome present more than twice a week
* Medical history of epilepsy
* Non stable psychiatric disorder
* Pregnancy, breastfeeding
* Subject deprived of liberty or protected by law (tutorship, curatorship).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of neurophysiological arousal response within 5 seconds after a subthreshold thermoalgic stimulation applied during parasomniac episodes. | within 5 seconds after stimulation

SECONDARY OUTCOMES:
Temperature of the thermoalgic stimulation during wakefulness associated with a nociceptive perception of 5/10 on a visual analogic scale | on inclusion
Minimal temperature of thermoalgic stimulations associated with a neurophysiological arousal response in NREM sleep stage 2 | within 5 seconds
Nociceptive behavioural response | within 5 seconds after a subthreshold thermoalgic stimulations applied during sleep and parasomniac episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France